CLINICAL TRIAL: NCT03233893
Title: Radiographic Assessment of Calcific Bridge Formation by Light Activated Calcium Silicate Versus Light Activated Calcium Hydroxide in Management of Simple Deeply Seated Carious Lesions With Partial Caries Removal
Brief Title: Radiographic Assessment of Calcific Bridge Formation by Light Activated Calcium Silicate Versus Calcium Hydroxide for Deep Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, basma gamal hassan, Resident of conservative department ,faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-07-21
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-07

CONDITIONS: Deep Carious Lesions
Keywords: based dentin substitute; dentin bridge; tertiary dentin; indirect pulp treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcome assessor will be blinded in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- light activated calcium silicate (Experimental): Apply light activated calcium silicate in deep occlusal caries lesions and taking the base line image for the first group after restoring the cavity with composite restoration and taking the follow up x-ray image after one year to measure the calcific bridge formation.
  Interventions: Other: light activated calcium silicate
- light activated calcium hydroxide (Active Comparator): Apply the light activated calcium hydroxide in deep occlusal carious lesions and taking the base line image for the second group after restoring with composite restoration and taking the follow up x-ray image after one year to measure the calcific bridge formation.
  Interventions: Other: light activated calcium silicate

INTERVENTIONS:
Other: light activated calcium silicate — for the first group light activated calcium silicate can be easily placed by a 20 second light cure and ability to be syringed directly on to the cavity preparation and restore the cavity by composite restoration.
  for the second group using light activated calcium hydroxide is placed by placing a disposable tip securely on to the syringe then light cure for 20 seconds depending on the light cure unit and restore the cavity with composite restoration.
  Other Names: light activated calcium hydroxide

SUMMARY:
sixty participants will be divided in to two groups (n=30) of patient treated by partial caries removal according to the capping material (A),where (A1)represents calcium silicate group,(A2)represent calcium hydroxide group.Apply light activated calcium silicate for group (A1) in deep occlusal caries and taking the base line image after restoring the cavity with composite restoration and apply light activated calcium hydroxide for(A2)group in deep occlusal caries and taking the base line image after restoring with composite restoration.Take follow up image after one year to measure the calcific bridge formation for both groups.

DETAILED DESCRIPTION:
Management of deep carious lesion may constitute a real challenge for the operator.The basic idea for treating deep caries is to enhance calcific reparative capacity.Calcium hydroxide has been the gold standard as a capping material but there are some drawbacks like solubility,gaps formation and mechanical instability so a need for a capping material such as calcium silicate has shown several advantages.

Sixty participants will be divided in to two groups (n=30) of patient treated by partial caries removal.The first group(A1) will be treated by light activated calcium silicate and the second group(A2) will be treated by light activated calcium hydroxide after partial caries removal of deep occlusal caries then restore by composite restoration.Paralleling technique using film holders and custom made bite blocks will be used to standardize the serial radiographs and to prevent the distortion of the radiographic image.An increase in dentin thickness will be measured through sequential imaging by soft ware named Digora (Digora Optime,Soredex,Helsinki,Finland) will be used for measurements by digitalizing the scanned image.All images will be studied carefully for an increase in dentin thickness keeping the reference point constant from the furcation area.

ELIGIBILITY:
Inclusion Criteria:

* Normal adults will be recruited in this study ,all the volunteers participated in this experiment will be healthy looking free medical history.
* Patients have simple deep carious lesions in his /her mouth with no pain or history of sensitivity to cold which disappear immediately after removal of the stimulus.

Exclusion Criteria:

* Medically compromised patients and teeth with history of spontaneous pain or tenderness to percussion were excluded from the study.
* Pregnant females will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
calcific bridge formation will be measured by digora software | 1 year
  in millimeters

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grewal N, Salhan R, Kaur N, Patel HB. Comparative evaluation of calcium silicate-based dentin substitute (Biodentine(R)) and calcium hydroxide (pulpdent) in the formation of reactive dentin bridge in regenerative pulpotomy of vital primary teeth: Triple blind, randomized clinical trial. Contemp Clin Dent. 2016 Oct-Dec;7(4):457-463. doi: 10.4103/0976-237X.194116. PMID 27994411
- See also: comparative evaluation of calcium silicate -based dentin substitute (Biodentine) and calcium hydroxide (pulpdent) in the formation of reactive dentin bridge in regenerative pulpotomy of vital primary teeth — http://www.contempclindent.org